CLINICAL TRIAL: NCT02953678
Title: A Single-Cohort, Phase 2 Study of Ruxolitinib in Combination With Corticosteroids for the Treatment of Steroid-Refractory Acute Graft-Versus-Host Disease (REACH-1)
Brief Title: A Study of Ruxolitinib in Combination With Corticosteroids for the Treatment of Steroid-Refractory Acute Graft-Versus-Host Disease (REACH-1)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Incyte Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: INCB 18424-271 (REACH-1)
Expanded Access: NCT03147742 (Approved for marketing)
Record Dates: First submitted 2016-11-01; First posted 2016-11-03 (Estimated); Results first posted 2019-08-20 (Actual); Last update posted 2021-11-24 (Actual); Status verified 2021-10

CONDITIONS: Graft-versus-host Disease (GVHD)
Keywords: Graft-versus-host disease (GVHD); acute GVHD; steroid-refractory; ruxolitinib; Janus kinase inhibitor
MeSH Terms: conditions — Graft vs Host Disease | interventions — ruxolitinib; Prednisone; Methylprednisolone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Ruxolitinib in combination with corticosteroids (Experimental): Participants began oral administration of ruxolitinib at 5 mg twice daily (BID); if stable after the first 3 days of treatment, the dose could be increased to 10 mg BID.
  Interventions: Drug: Ruxolitinib; Drug: Prednisone or methylprednisolone

INTERVENTIONS:
Drug: Ruxolitinib
  Other Names: Jakafi; INCB018424
Drug: Prednisone or methylprednisolone — Either oral prednisone or IV methylprednisolone may be used to begin corticosteroid treatment at the investigator's discretion.

SUMMARY:
The purpose of this study was to assess the efficacy of ruxolitinib in combination with corticosteroids in subjects with Grades II to IV steroid-refractory acute graft-versus-host disease (GVHD).

ELIGIBILITY:
Inclusion Criteria:

* Have undergone first allogeneic hematopoietic stem cell transplantation (allo-HSCT) from any donor source using bone marrow, peripheral blood stem cells, or cord blood for hematologic malignancies. Recipients of nonmyeloablative and myeloablative conditioning regimens are eligible.
* Clinically suspected Grades II to IV acute GVHD as per MAGIC guidelines, occurring after allo-HSCT with any conditioning regimen and any anti-GVHD prophylactic program.
* Subjects with steroid-refractory acute GVHD, defined as any of the following:

  * Subjects with progressive GVHD (ie, increase in stage in any organ system or any new organ involvement) after 3 days of primary treatment with methylprednisolone ≥ 2 mg/kg per day (or equivalent).
  * Subjects with GVHD that has not improved (ie, decrease in stage in at least 1 involved organ system) after 7 days of primary treatment with methylprednisolone ≥ 2 mg/kg per day (or equivalent).
  * Subjects who previously began corticosteroid therapy at a lower dose (at least 1 mg/kg per day methylprednisolone) but develop new GVHD in another organ system.
  * Subjects who cannot tolerate a corticosteroid taper, that is, begin corticosteroids at 2.0 mg/kg per day, demonstrate response, but progress before a 50% decrease from the initial starting dose of corticosteroids is achieved.
* Evidence of myeloid engraftment (eg, absolute neutrophil count ≥ 0.5 × 10^9/L for 3 consecutive days if ablative therapy was previously used). Use of growth factor supplementation is allowed.
* Be willing to avoid pregnancy or fathering children

Exclusion Criteria:

* Has received more than 1 allo-HSCT.
* Has received more than 1 systemic treatment in addition to corticosteroids for acute GVHD.
* Presence of GVHD overlap syndrome as per NIH guidelines.
* Subjects who have had a splenectomy.
* Presence of an active uncontrolled infection. An active uncontrolled infection is defined as hemodynamic instability attributable to sepsis or new symptoms, worsening physical signs, or radiographic findings attributable to infection. Persisting fever without signs or symptoms will not be interpreted as an active uncontrolled infection.
* Known human immunodeficiency virus infection.
* Active hepatitis B virus (HBV) or hepatitis C virus infection that requires treatment or at risk for HBV reactivation. Subjects whose immune status is unknown or uncertain must have results confirming immune status before enrollment.
* Serum creatinine > 2.0 mg/dL or creatinine clearance < 40 mL/min measured or calculated by Cockcroft-Gault equation.
* Subjects with evidence of relapsed primary disease, or subjects who have been treated for relapse after the allo-HSCT was performed.
* Unresolved toxicity or complications (other than acute GVHD) due to previous allo-HSCT.
* Any corticosteroid therapy for indications other than GVHD at doses of methylprednisolone or equivalent > 1 mg/kg per day within 7 days of enrollment.
* Severe organ dysfunction unrelated to underlying GVHD, including:

  * Cholestatic disorders or unresolved veno-occlusive disease of the liver (defined as persistent bilirubin abnormalities not attributable to GVHD and ongoing organ dysfunction).
  * Clinically significant or uncontrolled cardiac disease including unstable angina, acute myocardial infarction within 6 months from Day 1 of study drug administration, New York Heart Association Class III or IV congestive heart failure, circulatory collapse requiring vasopressor or inotropic support, or arrhythmia that requires therapy.
  * Clinically significant respiratory disease that requires mechanical ventilation support or 50% oxygen.
* Currently breast feeding.
* Received Janus kinase inhibitor (JAK) therapy after allo-HSCT for any indication. Treatment with a JAK inhibitor before allo-HSCT is permitted.
* Treatment with any other investigational agent, device, or procedure, within 21 days (or 5 half-lives, whichever is greater) of enrollment. Subjects participating in a GVHD prophylaxis study or conditioning regimen should be discussed with the sponsor's medical monitor before enrollment.
* Any condition that would, in the investigator's judgment, interfere with full participation in the study, including administration of study drug and attending required study visits; pose a significant risk to the subject; or interfere with interpretation of study data.
* Known allergies, hypersensitivity, or intolerance to any of the study medications, excipients, or similar compounds.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2016-12-30 (Actual); Primary Completion 2018-01-31 (Actual); Study Completion 2019-08-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Fitzroy Dawkins, MD, Study Director — Incyte Corporation
Locations (32):
- United States (32):
  - Tucson, Arizona
  - Duarte, California
  - La Jolla, California
  - Los Angeles, California
  - Stanford, California
  - Denver, Colorado
  - Gainesville, Florida
  - Miami, Florida
  - Tampa, Florida
  - Atlanta, Georgia
  - Chicago, Illinois
  - Lexington, Kentucky
  - Boston, Massachusetts
  - Grand Rapids, Michigan
  - Minneapolis, Minnesota
  - St Louis, Missouri
  - Hackensack, New Jersey
  - New York, New York
  - Rochester, New York
  - Charlotte, North Carolina
  - Cincinnati, Ohio
  - Cleveland, Ohio
  - Philadelphia, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Nashville, Tennessee
  - Dallas, Texas
  - San Antonio, Texas
  - Salt Lake City, Utah
  - Seattle, Washington
  - Morgantown, West Virginia
  - Madison, Wisconsin
  - Milwaukee, Wisconsin

REFERENCES:
- [Derived] Jagasia M, Perales MA, Schroeder MA, Ali H, Shah NN, Chen YB, Fazal S, Dawkins FW, Arbushites MC, Tian C, Connelly-Smith L, Howell MD, Khoury HJ. Ruxolitinib for the treatment of steroid-refractory acute GVHD (REACH1): a multicenter, open-label phase 2 trial. Blood. 2020 May 14;135(20):1739-1749. doi: 10.1182/blood.2020004823. PMID 32160294
- [Derived] Jagasia M, Zeiser R, Arbushites M, Delaite P, Gadbaw B, Bubnoff NV. Ruxolitinib for the treatment of patients with steroid-refractory GVHD: an introduction to the REACH trials. Immunotherapy. 2018 Apr;10(5):391-402. doi: 10.2217/imt-2017-0156. Epub 2018 Jan 10. PMID 29316837

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 26 study centers in the United States.
Groups:
- Ruxolitinib in Combination With Corticosteroids: Participants began oral administration of ruxolitinib at 5 mg twice a day (BID); if stable after the first 3 days of treatment, the dose may be increased to 10 mg BID. Participants did receive prednisone 2.5 mg/kg per day orally (PO) or methylprednisolone 2.0 mg/kg per day IV.
Period: Overall Study
Arm/Group | Ruxolitinib in Combination With Corticosteroids
Started | 71
Completed | 0
Not Completed | 71
Not completed — Adverse Event | 20
Not completed — Death | 7
Not completed — Physician Decision | 23
Not completed — Progressive Disease of GVHD | 7
Not completed — Relapse of Underlying Malignancy | 3
Not completed — Withdrawal by participant | 3
Not completed — Includes 2 participants who discontinued ruxolitinib treatment because of clinical improvement | 5
Not completed — Participants were transferred to commercial product. | 3

BASELINE CHARACTERISTICS:
Population: The efficacy evaluable population included all participants enrolled in the study.
Groups:
- Ruxolitinib in Combination With Corticosteroids: Participants began oral administration of ruxolitinib at 5 mg BID; if stable after the first 3 days of treatment, the dose may be increased to 10 mg BID. Participants did receive prednisone 2.5 mg/kg per day orally (PO) or methylprednisolone 2.0 mg/kg per day IV.
Arm/Group | Ruxolitinib in Combination With Corticosteroids
Number analyzed (Participants) | 71
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.9 (14.18)
Age, Customized [Count of Participants; unit: Participants]
  < 65 years | 58
  ≥ 65 years | 13
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36
  Male | 35
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9
  Not Hispanic or Latino | 60
  Unknown or Not Reported | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 66
  More than one race | 0
  Unknown or Not Reported | 0
Height [Mean (Standard Deviation); unit: cm] — Population: Height was not obtained for 5 participants.
  cm
    number analyzed (Participants) | 66
    (all) | 170.2 (10.64)
Weight [Mean (Standard Deviation); unit: kg] | 78.64 (21.651)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] — Population: Height was not obtained for 5 participants; BMI could not be calculated for these participants.
  kg/m^2
    number analyzed (Participants) | 66
    (all) | 26.83 (6.193)
Body Surface Area (BSA) [Mean (Standard Deviation); unit: m^2] — Population: Height was not obtained for 5 participants; BSA could not be calculated for these participants.
  m^2
    number analyzed (Participants) | 66
    (all) | 1.91 (0.301)
Eastern Cooperative Oncology Group (ECOG) grade at baseline [Count of Participants; unit: Participants] — ECOG scores are from 0-5: 0 = fully active, able to carry on all predisease performance without restriction; 1 = restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, eg, light house work, office work; 2 = ambulatory and capable of all self-care but unable to carry out any work activities, up and about more than 50% of waking hours; 3 = capable of only limited self-care, confined to bed or chair more than 50% of waking hours; 4 = completely disabled, cannot carry on any self-care, totally confined to bed or chair; and 5 = dead.
  Participants
    ECOG - 0 | 3
    ECOG - 1 | 24
    ECOG - 2 | 25
    ECOG - 3 | 17
    ECOG - 4 | 1
    ECOG - 5 | 0
    Missing | 1

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate (ORR) at Day 28
Description: Defined as the percentage of participants demonstrating a complete response (CR), very good partial response (VGPR), or partial response (PR).
Time Frame: From baseline to Day 28
Population: Efficacy Evaluable Participants who had a CR, VGPR, or PR at Day 28 response assessment or other response assessments within ± 2 days of Day 28, on or before the start of new anti-GVHD therapy
Measure: Count of Participants; unit: Participants
Arm/Group | Ruxolitinib in Combination With Corticosteroids
Number analyzed (Participants) | 71
Participants
  Responders - CR | 19
  Responders - VGPR | 7
  Responders - PR | 13
Statistical Analysis 1: Comparison: Ruxolitinib in Combination With Corticosteroids; Test type: Other; Exact method for binomial distributions = 54.9, 95% CI 2-sided [42.7 to 66.8]

2. Secondary Outcome: Overall Response Rate (ORR)
Description: Defined as the percentage of participants demonstrating a CR, VGPR, or PR.
Time Frame: From baseline to days 14, 56, and 100
Population: Efficacy Evaluable Population included all participants enrolled in this study.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Ruxolitinib in Combination With Corticosteroids: Participants began oral administration of ruxolitinib at 5 mg BID; if stable after the first 3 days of treatment, the dose may be increased to 10 mg BID up to approximately 27 months. Participants did receive prednisone daily orally (PO) daily or methylprednisolone daily intravenously( IV) as per protocol.
Arm/Group | Ruxolitinib in Combination With Corticosteroids
Number analyzed (Participants) | 71
percentage of participants
  Day 14 | 62.0 [49.7 to 73.2]
  Day 56 | 36.6 [25.5 to 48.9]
  Day 100 | 32.4 [21.8 to 44.5]

3. Secondary Outcome: Nonrelapse Mortality (NRM)
Description: Defined as the proportion of subjects who died due to causes other than malignancy relapse.
Time Frame: From baseline to Months 6, 9, 12, and 24
Population: Efficacy Evaluable Participants including all responders as of the data cutoff (02 JUL 2018).
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Ruxolitinib in Combination With Corticosteroids
Number analyzed (Participants) | 71
percentage of participants
  6 months | 44.4 [32.5 to 55.7]
  9 months | 48.2 [35.8 to 59.5]
  12 months | 52.9 [39.6 to 64.5]
  24 months | 64.8 [46.0 to 78.5]

4. Secondary Outcome: Percentage of Participants With Six-month Duration of Response (DOR)
Description: Defined as the time from first response until graft-versus-host disease (GVHD) progression or death. DOR was assessed when all participants who were on the study completed the Day 180 visit.
Time Frame: From Baseline up to 6 months
Population: Efficacy Evaluable Population included all participants enrolled in this study. Participants who achieved ORR were analyzed for this outcome measure.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Ruxolitinib in Combination With Corticosteroids
Number analyzed (Participants) | 40
percentage of participants | 68.2 [49.6 to 81.2]

5. Secondary Outcome: Percentage of Participants With Three-month DOR
Description: Defined as the time from first response until GVHD progression or death. DOR was assessed when all participants who were on the study completed the Day 84 visit.
Time Frame: From Baseline up to 3 months
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Ruxolitinib in Combination With Corticosteroids
Number analyzed (Participants) | 40
percentage of participants | 84.5 [68.7 to 92.7]

6. Secondary Outcome: Relapse Rate
Description: Defined as the percentage of participants whose underlying malignancy relapsed.
Time Frame: From Baseline until death, withdrawal of consent, or the end of the study, whichever occurs first (up to approximately 24 months)
Population: Efficacy Evaluable Population included all participants enrolled in this study.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Ruxolitinib in Combination With Corticosteroids
Number analyzed (Participants) | 71
percentage of participants | 7.0 [2.3 to 15.7]

7. Secondary Outcome: Relapse-related Mortality Rate
Description: Defined as the percentage of participants whose malignancy relapsed and had a fatal outcome.
Time Frame: as for outcome 6
Population: Efficacy Evaluable Population included all participants enrolled in this study.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Ruxolitinib in Combination With Corticosteroids
Number analyzed (Participants) | 71
percentage of participants | 5.6 [1.6 to 13.8]

8. Secondary Outcome: Failure-free Survival (FFS)
Description: Defined as the time from first dose of ruxolitinib to the earliest date that a participant died, had a relapse/progression of the underlying malignancy, required additional therapy for aGVHD, or demonstrated signs or symptoms of chronic graft-versus-host disease (cGVHD).
Time Frame: as for outcome 6
Population: Efficacy Evaluable Participants
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Ruxolitinib in Combination With Corticosteroids
Number analyzed (Participants) | 71
days | 85.0 [42.0 to 158.0]

9. Secondary Outcome: Overall Survival (OS)
Description: Defined as the time from study enrollment (first day of ruxolitinib treatment) to death due to any cause.
Time Frame: as for outcome 6
Population: Efficacy Evaluable Participants: Participants who had CR, VGPR, or PR on or before the start of new anti-GVHD therapy.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Ruxolitinib in Combination With Corticosteroids
Number analyzed (Participants) | 71
days | 232.0 [93.0 to 675.0]

10. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAES), Serious TEAEs, And Grade 3 or Higher TEAEs
Description: AE was any unfavorable and unintended sign, symptom, or disease temporally associated with use of medical treatment or procedure that may or may not be considered related to the medical treatment or procedure. Serious AE was any untoward medical occurrence that results in death; is life-threatening; requires inpatient hospitalization or prolongation of present hospitalization; results in persistent or significant disability/incapacity; is a congenital anomaly/birth defect or is a medically important event that may not be immediately life-threatening or result in death or hospitalization. TEAE was an AE that was reported for the first time, or worsening of a pre-existing event after the first dose of study drug (until 30 days after the last dose of study drug). Severity of AEs was described and graded using the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE version 4.03). Grade 3 and above would constitute a severe, life-threatening, or death event.
Time Frame: From signing the informed consent form up to 30-35 days after the last dose of study treatment (up to 24 months)
Population: Safety Evaluable Population included all participants enrolled in the study who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Ruxolitinib in Combination With Corticosteroids
Number analyzed (Participants) | 71
Participants
  TEAEs | 71
  Serious TEAEs | 59
  Grade 3 or Higher TEAEs | 69

ADVERSE EVENTS:
Time Frame: From signing the informed consent form up to 30-35 days after the last dose of study treatment (up to 24 months)
Description: The safety evaluable population includes all participants enrolled in the study who received at least 1 dose of study drug.
Arm/Group | Ruxolitinib in Combination With Corticosteroids
All-Cause Mortality (participants affected / at risk) | 46/71
Serious Adverse Events (participants affected / at risk) | 59/71
Other Adverse Events (participants affected / at risk) | 69/71
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ruxolitinib in Combination With Corticosteroids (N=71)
Anaemia (Blood and lymphatic system disorders) | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 1
Cardiac arrest (Cardiac disorders) | 1
Myocardial infarction (Cardiac disorders) | 2
Palpitations (Cardiac disorders) | 1
Pulseless electrical activity (Cardiac disorders) | 1
Supraventricular tachycardia (Cardiac disorders) | 1
Blindness (Eye disorders) | 1
Eye disorder (Eye disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Abdominal pain upper (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 3
Dysphagia (Gastrointestinal disorders) | 1
Gastritis (Gastrointestinal disorders) | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 2
Nausea (Gastrointestinal disorders) | 2
Pneumatosis intestinalis (Gastrointestinal disorders) | 4
Retroperitoneal haematoma (Gastrointestinal disorders) | 1
Small intestinal haemorrhage (Gastrointestinal disorders) | 1
Toothache (Gastrointestinal disorders) | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 2
Multiple organ dysfunction syndrome (General disorders) | 2
Pain (General disorders) | 1
Pyrexia (General disorders) | 8
Sudden death (General disorders) | 1
Cholecystitis acute (Hepatobiliary disorders) | 1
Hepatic failure (Hepatobiliary disorders) | 2
Venoocclusive liver disease (Hepatobiliary disorders) | 1
Acute graft versus host disease (Immune system disorders) | 1
Graft versus host disease in gastrointestinal tract (Immune system disorders) | 1
Graft versus host disease in liver (Immune system disorders) | 1
Bacteraemia (Infections and infestations) | 4
Bronchopulmonary aspergillosis (Infections and infestations) | 1
Candida infection (Infections and infestations) | 1
Cellulitis (Infections and infestations) | 1
Citrobacter infection (Infections and infestations) | 1
Cystitis (Infections and infestations) | 1
Cytomegalovirus viraemia (Infections and infestations) | 1
Device related infection (Infections and infestations) | 2
Enterococcal infection (Infections and infestations) | 1
Enterocolitis infectious (Infections and infestations) | 1
Escherichia urinary tract infection (Infections and infestations) | 1
Fungaemia (Infections and infestations) | 1
Hepatic infection fungal (Infections and infestations) | 1
Influenza (Infections and infestations) | 2
Klebsiella bacteraemia (Infections and infestations) | 1
Lung infection (Infections and infestations) | 5
Mycotic endophthalmitis (Infections and infestations) | 1
Peritonitis (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 5
Pneumonia bacterial (Infections and infestations) | 1
Pneumonia legionella (Infections and infestations) | 1
Respiratory syncytial virus infection (Infections and infestations) | 1
Sepsis (Infections and infestations) | 9
Septic shock (Infections and infestations) | 3
Sialoadenitis (Infections and infestations) | 1
Sinusitis (Infections and infestations) | 1
Staphylococcal bacteraemia (Infections and infestations) | 2
Staphylococcal infection (Infections and infestations) | 1
Staphylococcal sepsis (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Fall (Injury, poisoning and procedural complications) | 1
Hip fracture (Injury, poisoning and procedural complications) | 1
Road traffic accident (Injury, poisoning and procedural complications) | 1
Alanine aminotransferase increased (Investigations) | 1
Aspartate aminotransferase increased (Investigations) | 1
Neutrophil count decreased (Investigations) | 1
Platelet count decreased (Investigations) | 2
Failure to thrive (Metabolism and nutrition disorders) | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1
Hyponatraemia (Metabolism and nutrition disorders) | 2
Back pain (Musculoskeletal and connective tissue disorders) | 1
Groin pain (Musculoskeletal and connective tissue disorders) | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1
Acute myeloid leukaemia recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Encephalopathy (Nervous system disorders) | 1
Headache (Nervous system disorders) | 2
Confusional state (Psychiatric disorders) | 1
Mental status changes (Psychiatric disorders) | 3
Suicidal ideation (Psychiatric disorders) | 1
Acute kidney injury (Renal and urinary disorders) | 4
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 7
Deep vein thrombosis (Vascular disorders) | 1
Hypotension (Vascular disorders) | 2
Enterocolitis (Gastrointestinal disorders) | 1
Disease progression (General disorders) | 2
Fatigue (General disorders) | 1
Cholecystitis (Hepatobiliary disorders) | 1
Liver injury (Hepatobiliary disorders) | 1
Enterococcal sepsis (Infections and infestations) | 1
Vascular access complication (Injury, poisoning and procedural complications) | 1
Influenza like illness (General disorders) | 1
Upper respiratory tract infection (Infections and infestations) | 1
Syncope (Nervous system disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ruxolitinib in Combination With Corticosteroids (N=71)
Anaemia (Blood and lymphatic system disorders) | 45
Neutropenia (Blood and lymphatic system disorders) | 6
Thrombocytopenia (Blood and lymphatic system disorders) | 13
Pericardial effusion (Cardiac disorders) | 7
Sinus tachycardia (Cardiac disorders) | 14
Dry eye (Eye disorders) | 11
Vision blurred (Eye disorders) | 8
Abdominal distension (Gastrointestinal disorders) | 11
Abdominal pain (Gastrointestinal disorders) | 15
Ascites (Gastrointestinal disorders) | 6
Constipation (Gastrointestinal disorders) | 13
Diarrhoea (Gastrointestinal disorders) | 20
Dry mouth (Gastrointestinal disorders) | 11
Dyspepsia (Gastrointestinal disorders) | 5
Dysphagia (Gastrointestinal disorders) | 5
Flatulence (Gastrointestinal disorders) | 11
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 4
Haemorrhoids (Gastrointestinal disorders) | 7
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 10
Nausea (Gastrointestinal disorders) | 23
Stomatitis (Gastrointestinal disorders) | 5
Vomiting (Gastrointestinal disorders) | 16
Chills (General disorders) | 8
Fatigue (General disorders) | 22
Malaise (General disorders) | 6
Non-cardiac chest pain (General disorders) | 7
Oedema (General disorders) | 4
Oedema peripheral (General disorders) | 33
Pyrexia (General disorders) | 11
Hypogammaglobulinaemia (Immune system disorders) | 5
BK virus infection (Infections and infestations) | 5
Cytomegalovirus infection (Infections and infestations) | 9
Cytomegalovirus viraemia (Infections and infestations) | 4
Enterococcal infection (Infections and infestations) | 6
Staphylococcal infection (Infections and infestations) | 4
Urinary tract infection (Infections and infestations) | 6
Contusion (Injury, poisoning and procedural complications) | 5
Fall (Injury, poisoning and procedural complications) | 14
Alanine aminotransferase increased (Investigations) | 18
Aspartate aminotransferase increased (Investigations) | 17
Blood alkaline phosphatase increased (Investigations) | 9
Blood bilirubin increased (Investigations) | 11
Blood creatinine increased (Investigations) | 13
International normalised ratio increased (Investigations) | 7
Lymphocyte count decreased (Investigations) | 8
Neutrophil count decreased (Investigations) | 27
Platelet count decreased (Investigations) | 32
Weight decreased (Investigations) | 7
White blood cell count decreased (Investigations) | 21
Acidosis (Metabolism and nutrition disorders) | 6
Decreased appetite (Metabolism and nutrition disorders) | 16
Dehydration (Metabolism and nutrition disorders) | 5
Hyperglycaemia (Metabolism and nutrition disorders) | 17
Hyperkalaemia (Metabolism and nutrition disorders) | 8
Hypermagnesaemia (Metabolism and nutrition disorders) | 6
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 9
Hypoalbuminaemia (Metabolism and nutrition disorders) | 13
Hypocalcaemia (Metabolism and nutrition disorders) | 22
Hypoglycaemia (Metabolism and nutrition disorders) | 10
Hypokalaemia (Metabolism and nutrition disorders) | 34
Hypomagnesaemia (Metabolism and nutrition disorders) | 24
Hyponatraemia (Metabolism and nutrition disorders) | 13
Hypophosphataemia (Metabolism and nutrition disorders) | 19
Arthralgia (Musculoskeletal and connective tissue disorders) | 13
Back pain (Musculoskeletal and connective tissue disorders) | 16
Muscular weakness (Musculoskeletal and connective tissue disorders) | 24
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 4
Myalgia (Musculoskeletal and connective tissue disorders) | 5
Pain in extremity (Musculoskeletal and connective tissue disorders) | 12
Dizziness (Nervous system disorders) | 10
Dysgeusia (Nervous system disorders) | 4
Encephalopathy (Nervous system disorders) | 4
Headache (Nervous system disorders) | 13
Lethargy (Nervous system disorders) | 5
Paraesthesia (Nervous system disorders) | 4
Peripheral sensory neuropathy (Nervous system disorders) | 4
Somnolence (Nervous system disorders) | 6
Syncope (Nervous system disorders) | 4
Tremor (Nervous system disorders) | 7
Anxiety (Psychiatric disorders) | 10
Confusional state (Psychiatric disorders) | 9
Delirium (Psychiatric disorders) | 6
Depression (Psychiatric disorders) | 11
Hallucination (Psychiatric disorders) | 4
Insomnia (Psychiatric disorders) | 10
Acute kidney injury (Renal and urinary disorders) | 13
Haematuria (Renal and urinary disorders) | 12
Micturition urgency (Renal and urinary disorders) | 4
Pollakiuria (Renal and urinary disorders) | 10
Urinary incontinence (Renal and urinary disorders) | 6
Urinary retention (Renal and urinary disorders) | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 15
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 24
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 8
Hiccups (Respiratory, thoracic and mediastinal disorders) | 4
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 7
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 8
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 9
Productive cough (Respiratory, thoracic and mediastinal disorders) | 5
Dry skin (Skin and subcutaneous tissue disorders) | 7
Erythema (Skin and subcutaneous tissue disorders) | 4
Pruritus (Skin and subcutaneous tissue disorders) | 4
Rash (Skin and subcutaneous tissue disorders) | 6
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 9
Hypertension (Vascular disorders) | 16
Hypotension (Vascular disorders) | 14
Pain (General disorders) | 4
Upper Respiratory Tract Infection (Infections and infestations) | 6
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Following the first publication, the Institution and/or Principal Investigator may publish data or results from the Study, provided, however, that the Institution and/or Principal Investigator submits the proposed publication to the Sponsor for review at least sixty (60) days prior to the date of the proposed publication. Sponsor may remove from the proposed publication any information that is considered confidential and/or proprietary other than Study data and results.

DOCUMENTS (2):
  • Study Protocol (2016-10-04): https://cdn.clinicaltrials.gov/large-docs/78/NCT02953678/Prot_000.pdf
  • Statistical Analysis Plan (2017-07-24): https://cdn.clinicaltrials.gov/large-docs/78/NCT02953678/SAP_001.pdf